CLINICAL TRIAL: NCT00681499
Title: Long-term Evaluation of the Quality of Life After Major Hepatic Resection for Malignant and Benign Diseases.
Brief Title: Quality of Life After Liver Resection
Status: Completed | Type: Observational
Sponsor: University of Bern (Other)
Responsible Party: Vanessa Banz, MD, Dep. of Visceral and Transplant surgery, Bern University Hospital, Switzerland
Other Study IDs: KEK 18/08
Record Dates: First submitted 2008-05-19; First posted 2008-05-21 (Estimated); Last update posted 2015-11-13 (Estimated); Status verified 2015-11

CONDITIONS: Liver Diseases; Liver Neoplasms
Keywords: Quality of Life; Liver Neoplasms; Surgical procedures, Operative
MeSH Terms: conditions — Liver Diseases; Liver Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- malignant: eg. hepatocellular carcinoma, colorectal liver metastases
- benign: eg. liver cysts, traumatic liver injuries, adenoma etc

SUMMARY:
Patients with malignant diseases are increasingly receiving more extensive hepatic resections, with im-proved preoperative and postoperative care leading to a reduced postoperative morbidity and mortality. In this setting, postoperative quality of life may become as important as overall patient survival. In this study we will be investigating the effect of the initial disease for which hepatic resection was carried out on short- and long-term quality of life.

DETAILED DESCRIPTION:
Background: Due to advances in operative methods and perioperative care, mortality and morbidity following major hepatic resection have decreased substantially, making long-term quality of life (QoL) an increasingly prominent issue.

Objectives: We plan on evaluating whether postoperative diagnosis is associated with long-term QoL and health in patients who require hepatic surgery for benign or malignant diseases and how QoL evolves with time.

Method: QoL will be evaluated using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core-30 and the liver-specific QLQ-LMC21 module. All patients requiring hepatic surgery aged >18 years will be included in the study. QoL evaluation is carried out preoperatively and at set intervals postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Patients with planned liver resection

Exclusion Criteria

* Patients with biopsy of the liver only
* Inability of understanding the questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients requiring liver resection for any benign or malignant liver diseases, including secondary tumours
Sampling Method: Non-Probability Sample
Enrollment: 198 (Actual)
Dates: Start 2008-02; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Quality of Life | preoperatively, 1-,3-,6-,12 months postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Banz, MD, Principal Investigator — Dep. of Visceral and transplant Surgery, University Hospital Berne, Switzerland
Locations (1):
- Department of visceral and transplant surgery, Bern University Hospital, Bern, Switzerland

REFERENCES:
- [Background] Cella DF. Quality of life: concepts and definition. J Pain Symptom Manage. 1994 Apr;9(3):186-92. doi: 10.1016/0885-3924(94)90129-5. PMID 8014530
- [Background] Slevin ML. Quality of life: philosophical question or clinical reality? BMJ. 1992 Aug 22;305(6851):466-9. doi: 10.1136/bmj.305.6851.466. No abstract available. PMID 1392964
- [Background] Aaronson NK, Ahmedzai S, Bergman B, Bullinger M, Cull A, Duez NJ, Filiberti A, Flechtner H, Fleishman SB, de Haes JC, et al. The European Organization for Research and Treatment of Cancer QLQ-C30: a quality-of-life instrument for use in international clinical trials in oncology. J Natl Cancer Inst. 1993 Mar 3;85(5):365-76. doi: 10.1093/jnci/85.5.365. PMID 8433390
- [Background] Kavadas V, Blazeby JM, Conroy T, Sezer O, Holzner B, Koller M, Buckels J; EORTC Quality of Life Group. Development of an EORTC disease-specific quality of life questionnaire for use in patients with liver metastases from colorectal cancer. Eur J Cancer. 2003 Jun;39(9):1259-63. doi: 10.1016/s0959-8049(03)00236-3. PMID 12763214
- [Background] Sloan JA, Loprinzi CL, Kuross SA, Miser AW, O'Fallon JR, Mahoney MR, Heid IM, Bretscher ME, Vaught NL. Randomized comparison of four tools measuring overall quality of life in patients with advanced cancer. J Clin Oncol. 1998 Nov;16(11):3662-73. doi: 10.1200/JCO.1998.16.11.3662. PMID 9817289
- [Background] Glimelius B, Hoffman K, Graf W, Pahlman L, Sjoden PO. Quality of life during chemotherapy in patients with symptomatic advanced colorectal cancer. The Nordic Gastrointestinal Tumor Adjuvant Therapy Group. Cancer. 1994 Feb 1;73(3):556-62. doi: 10.1002/1097-0142(19940201)73:33.0.co;2-8. PMID 8299077
- [Background] Sterkenburg CA, King B, Woodward CA. A reliability and validity study of the McMaster Quality of Life Scale (MQLS) for a palliative population. J Palliat Care. 1996 Spring;12(1):18-25. PMID 8857243
- [Background] Brunelli C, Costantini M, Di Giulio P, Gallucci M, Fusco F, Miccinesi G, Paci E, Peruselli C, Morino P, Piazza M, Tamburini M, Toscani F. Quality-of-life evaluation: when do terminal cancer patients and health-care providers agree? J Pain Symptom Manage. 1998 Mar;15(3):151-8. doi: 10.1016/s0885-3924(97)00351-5. PMID 9564116
- [Background] Tamames S, De Vega DS, Tamames S Jr. Surgical management of malignant tumors of the esophagogastric junction: a retrospective review of 188 patients. Int Surg. 1990 Apr-Jun;75(2):89-92. PMID 2379996
- [Background] Martin RC, Eid S, Scoggins CR, McMasters KM. Health-related quality of life: return to baseline after major and minor liver resection. Surgery. 2007 Nov;142(5):676-84. doi: 10.1016/j.surg.2007.04.026. PMID 17981187
- [Background] Chen L, Liu Y, Li GG, Tao SF, Xu Y, Tian H. Quality of life in patients with liver cancer after operation: a 2-year follow-up study. Hepatobiliary Pancreat Dis Int. 2004 Nov;3(4):530-3. PMID 15567739